CLINICAL TRIAL: NCT01574248
Title: Effect of Bradykinin Receptor Antagonism on ACE Inhibitor-associated Angioedema - a Mulitcenter Trial
Brief Title: Effect of Bradykinin Receptor Antagonism on ACE Inhibitor-associated Angioedema
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMC recommended discontinuation for futility and feasibility
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Nancy J. Brown, Chair Department of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000626
Record Dates: First submitted 2011-12-14; First posted 2012-04-10 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: ACE Inhibitor-associated Angioedema
Keywords: ACE inhibitor; Angioedema; Bradykinin; Swelling
MeSH Terms: conditions — Angioedema | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- icatibant (Experimental): 30 mg icatibant will be administered subcutaneously 0 and 6 hours after randomization
  Interventions: Drug: icatibant
- Placebo (Placebo Comparator): Subcutaneous at time 0 and 6 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: icatibant — Subcutaneous at time 0 and 6 hours
  Other Names: Firazyr; HOE140
  Arms: icatibant
Other: Placebo — Subcutaneous at time 0 and 6 hours
  Arms: Placebo

SUMMARY:
Individuals with heart disease or high blood pressure are often prescribed angiotensin converting enzyme (ACE) inhibitors to treat their disease. However, the use of ACE inhibitors can be associated with angioedema, a rare but life-threatening condition that causes swelling of the face and other body parts. This study will evaluate the effectiveness of the drug HOE-140 at decreasing symptoms of angioedema in people taking ACE inhibitors who develop the condition.

DETAILED DESCRIPTION:
People who take ACE inhibitors may develop angioedema, a condition that causes itchy and painful swelling beneath the skin around the eyes, lips, tongue, throat, hands, or feet. In severe cases, the throat may swell, obstructing the airway and leading to breathing difficulty. ACE inhibitors prevent the breakdown of a natural chemical in the body called bradykinin. Increased levels of bradykinin, which can cause swelling, may contribute to the development of angioedema. Blocking bradykinin receptor cells prevents bradykinin from initiating swelling and may lead to a possible decrease in angioedema symptoms. The purpose of this study is to evaluate the effectiveness of HOE-140, a bradykinin receptor blocker, at reducing symptoms in people with ACE inhibitor-associated angioedema.

This study will enroll people admitted to the emergency room or hospital who have a severe case of ACE inhibitor-associated angioedema. Participants will be randomly assigned to receive an injection of either HOE-140 or placebo. Initially, participants will undergo an electrocardiogram to measure the electrical activity of the heart. Then blood pressure measurements, blood collection, a physical exam to determine the extent and duration of swelling, and photographs of the swelling will occur at 2, 4, 8, 16, and 24 hours following the start of treatment. Questionnaires will be completed by study staff and participants to assess changes in angioedema symptoms and the extent of swelling. Participants will remain in the hospital for 24 to 48 hours, depending on the severity of their symptoms. Blood will be collected at a follow-up visit that will occur 7 days after the resolution of angioedema symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The subject has ongoing angioedema while taking an ACE inhibitor.
* The subject is between 18 and 80 years of age.

Exclusion Criteria:

* The subject has had angioedema while not taking an ACE inhibitor.
* The subject's angioedema only involves the bowel.
* The subject is known to be pregnant or has a positive urine pregnancy test.
* The subject has started on an oral contraceptive within the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Brown, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Byrd JB, Adam A, Brown NJ. Angiotensin-converting enzyme inhibitor-associated angioedema. Immunol Allergy Clin North Am. 2006 Nov;26(4):725-37. doi: 10.1016/j.iac.2006.08.001. PMID 17085287
- [Background] Brown NJ, Ray WA, Snowden M, Griffin MR. Black Americans have an increased rate of angiotensin converting enzyme inhibitor-associated angioedema. Clin Pharmacol Ther. 1996 Jul;60(1):8-13. doi: 10.1016/S0009-9236(96)90161-7. PMID 8689816
- [Background] Brown NJ, Byiers S, Carr D, Maldonado M, Warner BA. Dipeptidyl peptidase-IV inhibitor use associated with increased risk of ACE inhibitor-associated angioedema. Hypertension. 2009 Sep;54(3):516-23. doi: 10.1161/HYPERTENSIONAHA.109.134197. Epub 2009 Jul 6. PMID 19581505
- [Background] Gainer JV, Morrow JD, Loveland A, King DJ, Brown NJ. Effect of bradykinin-receptor blockade on the response to angiotensin-converting-enzyme inhibitor in normotensive and hypertensive subjects. N Engl J Med. 1998 Oct 29;339(18):1285-92. doi: 10.1056/NEJM199810293391804. PMID 9791144
- [Background] Zuraw BL. Clinical practice. Hereditary angioedema. N Engl J Med. 2008 Sep 4;359(10):1027-36. doi: 10.1056/NEJMcp0803977. No abstract available. PMID 18768946
- [Background] Verresen L, Fink E, Lemke HD, Vanrenterghem Y. Bradykinin is a mediator of anaphylactoid reactions during hemodialysis with AN69 membranes. Kidney Int. 1994 May;45(5):1497-503. doi: 10.1038/ki.1994.195. PMID 8072263
- [Background] Krieter DH, Grude M, Lemke HD, Fink E, Bonner G, Scholkens BA, Schulz E, Muller GA. Anaphylactoid reactions during hemodialysis in sheep are ACE inhibitor dose-dependent and mediated by bradykinin. Kidney Int. 1998 Apr;53(4):1026-35. doi: 10.1111/j.1523-1755.1998.00837.x. PMID 9551414
- [Background] Bork K, Frank J, Grundt B, Schlattmann P, Nussberger J, Kreuz W. Treatment of acute edema attacks in hereditary angioedema with a bradykinin receptor-2 antagonist (Icatibant). J Allergy Clin Immunol. 2007 Jun;119(6):1497-503. doi: 10.1016/j.jaci.2007.02.012. Epub 2007 Apr 5. PMID 17418383
- [Background] Brown NJ, Snowden M, Griffin MR. Recurrent angiotensin-converting enzyme inhibitor--associated angioedema. JAMA. 1997 Jul 16;278(3):232-3. doi: 10.1001/jama.278.3.232. PMID 9218671

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Icatibant | Placebo
Started | 15 | 18
Completed | 12 | 18
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Missing primary endpoint data | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Icatibant | Placebo | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.4) | 60.7 (10.8) | 58.9 (11.8)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Angioedema
Description: Time interval between initiation of treatment and when there is no symptom, by visual analog scale <1 cm. Data provided are for worst symptom.
Time Frame: 48 hours
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
hours | 36 [24 to 48] | 24 [6 to 48]

2. Secondary Outcome: Number of Participants With Admission to Intensive Care Unit
Time Frame: T0 to T48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
Participants | 6 | 6

3. Secondary Outcome: Number of Participants With Requirement for Intubation
Time Frame: T0 to T48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
Participants | 2 | 1

4. Secondary Outcome: Number of Participants Given Steroids
Time Frame: T0 to T48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
Participants | 11 | 16

5. Secondary Outcome: Number of Participants Given Histamine Receptor Type 1 (H1) and Type 2 (H2) Blockers
Time Frame: T0 to T48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
Participants | 11 | 16

6. Secondary Outcome: Number of Participants Given Epinephrine
Time Frame: T0 to T48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
Participants | 0 | 3

7. Secondary Outcome: Systolic Blood Pressure
Description: Average of blood pressure measurements from zero to forty-eight hours provided.
Time Frame: T0 to T48 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 12 | 18
mmHg | 134 (13) | 133 (17)

ADVERSE EVENTS:
Arm/Group | Icatibant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 1/12 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant (N=12) | Placebo (N=18)
low sperm count (Reproductive system and breast disorders) | 0 (0) | 1 (1)
elevated troponin (Cardiac disorders) | 0 (0) | 1 (1)
leukocytosis (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No